CLINICAL TRIAL: NCT02625935
Title: A Prospective Observational Study Evaluating Treatment Decision Impact of Prosigna® in Early Stage Breast Cancer Patients Who Are Candidates for Genomic Testing
Brief Title: Prospective Observational Study Evaluating Treatment Decision Impact of Prosigna® in Early Stage Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: NanoString Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-10140
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: Prosigna; estrogen receptor positive; node negative; HER2 negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE breast tumor tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This multicenter, prospectively designed study examines whether the Prosigna score influences physician and patient adjuvant treatment selection over and above currently used prognostic factors. This study also examines the impact of the test results on patients' reported outcomes, including their decisional conflict status and anxiety levels.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the extent to which the Prosigna test results affect the medical oncologist's treatment recommendations regarding adjuvant chemotherapy and actual treatments received for patients with early stage breast cancer conventionally considered candidates for genomic testing based on current treatment guidelines. The oncologist's initial recommendations will be based on the utilization of tools or algorithms based on clinical and pathologic factors. No genomic tools will be used in the initial assessment. Changes in recommendation after availability of Prosigna test results will include (1) hormonal therapy alone or (2) hormonal therapy plus chemotherapy, and (3) changes in types of chemotherapy if chemotherapy was recommended before and after the test.

ELIGIBILITY:
Inclusion Criteria:

* Surgically resected node-negative, estrogen receptor-positive, HER2-negative early-stage invasive breast cancer (T1-T2, N0, pN0 (i+), pN0 (mol+), M0)

  1. Estrogen receptor status will be evaluated by Immunohistochemistry (IHC) and more than 1% of stained tumor cells will be considered positive.
  2. HER2 status will be evaluated by IHC and/or by in-situ fluorescence hybridization (0 or 1+, or 2+ will be considered negative in the absence of in-situ fluorescence hybridization).
* Postmenopausal females, which is defined as:

  1. Natural Amenorrhea > 12 months, regardless of age
  2. Bilateral oophorectomy, regardless of age (the oophorectomy must have been carried out at least 4 weeks before entering the study)
  3. Radiological castration with amenorrhea > 3 months, regardless of age
  4. Hysterectomy and postmenopausal blood levels of FSH/LH
* Able to give informed consent
* Eligible for treatment of breast cancer with adjuvant chemotherapy, as determined by the treating physician
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Tumor specimen from core needle biopsy (CNB)
* Tumor stage T3-T4
* Non-invasive breast cancer (e.g., Paget's disease, DCIS)
* Tumors with nodes that are not N0, pN0 (i+), or pN0 (mol+)
* Tumors that are estrogen receptor (ER) negative or HER2-positive
* Have metastatic disease
* Have received another genomic test for prognosis of early breast cancer (i.e., Oncotype Dx, Mammaprint, or BCI)
* Unable to give informed consent
* Unable to complete patient reported outcome surveys
* Have contraindications for adjuvant chemotherapy, as determined by the treating physician

  o Age, performance status, significant comorbidities, etc.
* ECOG performance status > 1

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with node-negative, estrogen-receptor positive, HER2-negative early-stage breast cancer.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients for whom the choice of treatment was changed as a result of receiving the Prosigna test results. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Vacirca, MD, Principal Investigator — North Shore Hematology Oncology Associates
Locations (4):
- United States (4):
  - Florida Cancer Center, Fort Myers, Florida
  - New England Cancer Specialists, Scarborough, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - North Shore Hematology Oncology Assoaciates, East Setauket, New York